CLINICAL TRIAL: NCT00749983
Title: Effects of Creatine Supplementation in Women With Knee Osteoarthritis and Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0849/07
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Knee Osteoarthritis; Fibromyalgia
MeSH Terms: conditions — Osteoarthritis, Knee; Fibromyalgia | interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): creatine intake
  Interventions: Dietary Supplement: Creatine supplementation
- 2 (Placebo Comparator): placebo (dextrose) intake
  Interventions: Dietary Supplement: Dextrose supplementation

INTERVENTIONS:
Dietary Supplement: Creatine supplementation
  Arms: 1
Dietary Supplement: Dextrose supplementation
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether creatine associated or not to exercise training can improve physical performance in patients with knee osteoarthritis and fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill ACR criteria of knee osteoarthritis
* Fulfill ACR criteria of fibromyalgia

Exclusion Criteria:

* Athletes
* Drugs stable for at least three months before entering the study
* No limitations to resistance training

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Physical function | 12 weeks
  Assessed by the timed-stands test

SECONDARY OUTCOMES:
Strength | 12 weeks
  Assessed by the 1-repetition maximum test
Quality of life | 12 weeks
  health-related questionaires
Body composition | 12 weeks
  Assessed by DXA
Renal function | 12 weeks
  Assessed by 51Cr-EDTA

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo School of Medicine, São Paulo, São Paulo, Brazil